CLINICAL TRIAL: NCT06522503
Title: The Effect of a Stress Ball on Perceived Stress, Pain and Satisfaction in Cancer Patients: A Distraction-Based Intervention
Brief Title: Effect of Stress Ball on Perceived Stress, Pain and Satisfaction in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Aysegul Celik, Asst. Prof., RN, MSc, PhD, Izmir Bakircay University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: SB
Record Dates: First submitted 2024-07-12; First posted 2024-07-26 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Cancer
Keywords: cancer patient; perceived stress; pain; patient satisfaction
MeSH Terms: conditions — Neoplasms; Pain; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental)
  Interventions: Behavioral: stress ball
- control (No Intervention)

INTERVENTIONS:
Behavioral: stress ball — The intervention group was provided with a stress ball to be held in both hands for a period of five minutes prior to the insertion of the port catheter needle. They were instructed to squeeze the ball in their hands at regular intervals until the conclusion of the procedure.
  Arms: intervention

SUMMARY:
The objective of this study was to ascertain the impact of stress ball utilisation on perceived stress, pain and satisfaction levels during port catheter intervention in cancer patients. In this study, which was conducted in a randomised controlled design, a control group of cancer patients receiving chemotherapy (n=37) was assigned to receive standard care during port catheter needle insertion. An intervention group (n=37) was also formed, comprising patients who received stress ball application in addition to standard care. The intervention group was provided with a stress ball in both hands five minutes prior to the insertion of the port catheter needle and instructed to squeeze the ball in their hands at regular intervals until the conclusion of the procedure. Prior to the application, the descriptive characteristics of both groups were ascertained, and their perceived stress levels were assessed. Subsequently, the pain and perceived stress levels of both groups were documented. Additionally, the satisfaction levels of the intervention group regarding the stress ball application were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Diagnosed with cancer
* Undergoing active chemotherapy
* Willing to participate in the research .

Exclusion Criteria:

* Communication difficulties
* Complaints of peripheral neuropathy
* Refusal to participate in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
perceived stress level | baseline and end of the port catheterisation procedure (mean time 10 minutes)
  Perceived Stress Scale: The Perceived Stress Scale, comprising a total of 14 items, has been developed to assess the degree to which an individual perceives specific circumstances in their life as stressful. The scale is a 5-point Likert-type scale, with each item ranging from "Never (0)" to "Very often (4)". The total score obtained from the scale is indicative of the individual's stress level.

SECONDARY OUTCOMES:
pain level | End of the port catheterisation procedure (mean time 10 minutes)
  The Visual Analogue Scale (VAS): The Visual Analogue Scale is a frequently employed instrument for the assessment of pain intensity. It is a unidimensional scale with a length of 0-10 cm. The scale is anchored at 0 cm, which is defined as no pain, and 10 cm, which is defined as unbearable pain. As the score obtained from the scale increases, the pain intensity also increases.

OTHER OUTCOMES:
patient satisfaction level | End of the port catheterisation procedure (mean time 10 minutes)
  Visual Analog Scale-Satisfaction Level (VAS): The Visual Analogue Scale (VAS), comprising a 10-cm line, represents a valid and reliable instrument for measuring subjective emotions such as mood. In this study, a visual analogue scale (VAS) was employed as a means of evaluating patient satisfaction levels.

CONTACTS AND LOCATIONS:
Overall Officials: Aslıhan Öztürk Çetin, MSc, Study Chair — Izmir Bakircay University
Locations (1):
- Ayşegül Çelik, Izmir, Menemen, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No